CLINICAL TRIAL: NCT00250744
Title: Comparison of Aprepitant vs. Gabapentin in the Prevention of Delayed Nausea and Vomiting
Brief Title: Comparison of Aprepitant Versus Gabapentin in the Prevention of Delayed Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INST 3204C
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2009-12

CONDITIONS: Cancer
Keywords: delayed nausea and vomiting; Emetogenic Chemotherapy; Pilot Trial
MeSH Terms: conditions — Neoplasms; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Aprepitant vs. Gabapentin
- Arm B (Active Comparator)
  Interventions: Drug: Aprepitant vs. Gabapentin

INTERVENTIONS:
Drug: Aprepitant vs. Gabapentin — Gabapentin 300mg PO QHS day -2; 300mg PO BID day -1; 300mg PO TID days 0 through +5.
  Arms: Arm A
Drug: Aprepitant vs. Gabapentin — Aprepitant 125mg PO 60 minutes prior to chemotherapy on day 0; 80 mg PO QAM on days +1 and +2.
  Arms: Arm B

SUMMARY:
1. To compare the effectiveness of gabapentin (titrated to300mg TID days -2 to 5) with aprepitant (125mg on day 1 and 80mg on days 2 and 3) in the control of delayed nausea and vomiting associated with level 3, 4 or 5 emetogenic chemotherapy in patients who experienced delayed nausea and/or vomiting during their first cycle of chemotherapy.
2. To evaluate and compare the safety profile associated with each anti-emetic regimen.
3. To assess subject satisfaction with anti-emetic therapy.

DETAILED DESCRIPTION:
The purpose of study is to compare the effectiveness of aprepitant and gabapentin in treating "delayed" (days later) nausea and/or vomiting for patients receiving chemotherapy treatment for cancer. Patients on the study will receive aprepitant or gabapentin in addition to the standard medications used to prevent nausea and vomiting. Aprepitant is approved by the FDA for nausea and vomiting. Gabapentin is approved by the FDA for the treatment of seizures but it may be effective in controlling nausea and vomiting due to chemotherapy. Subjects receiving aprepitant will be receiving a proven treatment for delayed nausea and vomiting, while subjects receiving gabapentin will be receiving a drug that has only shown limited effectiveness.

Patients are eligible for participation in this study because they are going to receive chemotherapy that may cause nausea or vomiting. If patients have delayed nausea or vomiting after the first cycle of treatment, they will be offered a chance to receive additional treatments with their second cycle of chemotherapy. The University of New Mexico Health Sciences Center is sponsoring the study.

The first 40 patients enrolled in the study will participate in the pilot phase of the study. A pilot study is a smaller version of a full study to determine how effective the treatments are. All 40 patients in the pilot phase of the study will come from UNM. If the pilot phase is found to be successful, then the study will continue and approximately 200 patients will eventually be enrolled. The full study will be conducted at the University of New Mexico Cancer Research and Treatment Center (UNM CRTC), the New Mexico VA Healthcare System, and at members of the New Mexico Cancer Care Alliance.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients, 18 years of age or older, who are eligible for chemotherapy may participate in the trial if the following criteria are met:

1. Patients must have a diagnosis of malignant disease and be scheduled to receive single-day intravenous chemotherapy drug or combination of drugs that are considered to elicit level 3, 4 or 5 emesis (appendix A).
2. Males must be surgically sterilized, or agree to practice adequate contraceptive precautions during the study.
3. Females of non-childbearing potential (i.e. those who have been surgically sterilized, or who are at least one-year post menopausal) may enter the study. Females of childbearing potential must have a negative pregnancy test (urine or serum hCG) before entry into the study, and must agree to practice adequate contraceptive precautions during the study.
4. Written informed consent must be obtained before initiating any protocol specified procedures.

Exclusion Criteria:

Patients with any of the following are not eligible for enrollment in the study.

1. Any unstable medical disorder.
2. Participation in any drug trial in which the patient received an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the screening phase of this study.
3. Patients with serum creatinine ≥ 2 dL/mL; bilirubin ≥ 3 times ULN; or those with an ECOG performance status ≥ 3.
4. Patients with severe hepatic insufficiency as evidenced by ascites, encephalopathy, coagulopathy, or jaundice.
5. Patients prescribed corticosteroids except for replacement or maintenance doses up to 10mg prednisone or equivalent. Dexamethasone is permitted as a prophylactic component of the pre- and post-chemotherapy anti-emetic regimen as defined in this protocol.
6. Primary or secondary (from metastatic disease) brain neoplasm with:

   * Signs or symptoms of increased intracranial pressure or
   * Patients with brain metastases requiring treatment within 30 days of entry into the study.

   Signs or symptoms of cerebral edema will exclude a patient from entry into the study. Patients with symptomatically "silent" metastases may be enrolled into the study.
7. Patients who are known to be hypersensitive to gabapentin, any neurokinin-1 or dopamine receptor antagonist, 5-HT3 receptor antagonists, or corticosteroids.
8. Patients who are unwilling or unable to comply with the protocol.
9. Patients are excluded if they are receiving radiation therapy to any abdominal field (T10-L5) within 24 hours before the dose of study medication is given or if they are scheduled to receive such radiation during the period of assessment (study days 0-2 for arm A and study days 0-6 for arm B). Radiation to other fields is acceptable (e.g. pelvic radiation, thoracic radiation).
10. Patients who have had any nausea within one hour and/or emesis (vomiting and/or retching) within 24 hours before dosing of study medication.
11. Patients who have taken either gabapentin or aprepitant within four weeks of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To compare the effectiveness of gabapentin with aprepitant in the control of delayed nausea & vomiting associated with level 3, 4 or 5 emetogenic chemotherapy in pts who experienced delayed nausea and/or vomiting during their first cycle of chemotherapy. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Cheshire, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States